CLINICAL TRIAL: NCT01874730
Title: KOREAN Enhanced RecOvery Strategy for Colorectal Surgery
Acronym: KEROS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very slow accrual because sites have few open colorectal surgery
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00038567
Record Dates: First submitted 2013-06-04; First posted 2013-06-11 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Goal-oriented Fluid Therapy; Colorectal Surgery
Keywords: colorectal surgery; fluid therapy
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (SOC) (Other): Intraoperative fluid management includes Volulyte® (6% hydroxyethyl starch {HES} 130/0.4 in balanced solution) as the only colloid solution to be used, the daily dosage of Volulyte® is restricted to 50 ml/kg. Intraoperative anesthesia and postoperative analgesia will follow the established practice of the individual institution.
  Interventions: Drug: Volulyte® (6% HES 130/0.4 in balanced solution)
- Enhanced Recovery Strategy (ERS) group (Active Comparator): GDFT regimen using Volulyte® (6% HES 130/0.4 in balanced solution) during surgery. The daily dosage of Volulyte® is restricted to 50 ml/kg. Combined epidural-general anesthesia (CEGA) will be used intraoperatively and patient-controlled epidural analgesia (PCEA) will be used postoperatively in a multimodal analgesic regimen.
  Interventions: Other: Combined epidural-general anesthesia (CEGA); Drug: Volulyte® (6% HES 130/0.4 in balanced solution); Other: Patient-Controlled Epidural Analgesia (PCEA)

INTERVENTIONS:
Other: Combined epidural-general anesthesia (CEGA) — Combined epidural-general anesthesia (CEGA) will be used intraoperatively and patient-controlled epidural analgesia (PCEA) will be used postoperatively in a multimodal analgesic regimen.
  Arms: Enhanced Recovery Strategy (ERS) group
Drug: Volulyte® (6% HES 130/0.4 in balanced solution) — For the SOC Group: Intraoperative fluid management includes Volulyte® (6% HES 130/0.4 in balanced solution) as the only colloid solution to be used, the daily dosage of Volulyte® is restricted to 50 ml/kg.
  For the ERS Group:
  GDFT regimen will be utilized using Volulyte® (6% HES 130/0.4 in balanced solution) during surgery. The daily dosage of Volulyte® is restricted to 50 ml/kg.
Other: Patient-Controlled Epidural Analgesia (PCEA) — For the ERS Group, patient-controlled epidural analgesia (PCEA) will be used postoperatively in a multimodal analgesic regimen.
  Arms: Enhanced Recovery Strategy (ERS) group

SUMMARY:
This is a multi-centre study to take place in approximately 3 centers in Seoul, South Korea. The study will be carried out as a prospective, randomized, controlled, multicenter, clinical trial in patients undergoing colorectal surgery. The purpose of this study is to determine if an enhanced recovery strategy paying close attention to the type and amount of fluid given during the surgery with proper monitoring combined with a comprehensive perioperative pain management will have a better post-operative outcome compared to institutional standard of care (SOC), in patients undergoing surgery of the colon. One of the fluids used, Volulyte®, is an intravenous solution used to treat low blood volume. The Volulyte® solution being used in the study and the monitor used are approved by the Korean Food and Drug Administration

ELIGIBILITY:
Inclusion Criteria:

1. Elective, open colorectal surgery including sigmoid resections, i.e. with an upper rectal anastomosis and with or without planned stoma. If the planned surgery is a combined procedure, the associated procedure should not add more than 1 hour to the surgery time of the primary colorectal surgical procedure alone.
2. Both genders; age ≥ 45 years and ≤ 80 years.
3. ASA Grades I-III
4. Voluntary participation and signing the informed consent form

Exclusion Criteria:

1. Fluid overload (hyperhydration), especially in cases of pulmonary edema and congestive heart failure, or patients with severe cardiovascular disorders (New York Heart Association, NYHA III-IV)
2. Patients with significant cardiac arrhythmias or depending on pacemaker
3. Patients with impaired liver and/or kidney functions (ALT more than 2 times the normal upper limit and/or Serum Creatinine (SCr) more than 2 times the normal upper limit)
4. Renal failure with oliguria or anuria not related to hypovolemia
5. Patients receiving dialysis treatment
6. Patients with non-resectable malignancies
7. Patients who are non-cooperative or non-communicable
8. Patients with significant preoperative coagulation abnormalities
9. Patients receiving treatment with opioids for significant chronic pain
10. Patients in need of organ transplantation
11. Intracranial hemorrhage
12. Severe hypernatremia (Na+ > 155 mmol/l) or severe hyperchloremia (Cl- > 125 mmol/l)
13. Known hypersensitivity to hydroxyethyl starches
14. Participation in a clinical trial of an investigational drug or device within 30 days before study screening visit or is scheduled to receive an investigational product while participating in this study
15. Patients with evidenced bowel obstruction symptoms.
16. Contraindication to epidural anesthesia
17. Known pregnancy and lactation

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Postoperative Outcome | From Day 1 after surgery and duration of hospital stay (approximately 6 days after surgery)
  Postoperative outcome is defined as the number of patients who develop at least one postoperative complication during their hospital stay

SECONDARY OUTCOMES:
Postoperative outcome for each patient at postoperative day (POD) 30 | From Hospital Discharge (approximately 6 days after surgery), up to 4 weeks after day of surgery
  Postoperative outcome for each patient at postoperative day (POD) 30 is defined as whether the patient encountered at least one postoperative complication up to POD 30
Number of postoperative complications per group | Participants will be followed for the duration of hospital stay (approximately 6 days after surgery), and until 4 weeks from day of surgery
  Number of postoperative complications per group evaluated postoperatively from date of surgery, each hospital day, (post-operative days 1 through 5), at discharge from the hospital until 30 days from day of surgery.
Time to "clinically fit for discharge from hospital" | From 4 days after surgery to Hospital discharge (approximately 6 days after surgery)
  Time to "clinically fit for discharge from hospital" when defined discharge criteria are met (evaluation starts from POD 4 at 10 am each day till discharge).
Change in Postoperative pain | 1h, 2 h, 6 h, 24 h post-surgery, and post-operative days 1 through 5, and at discharge
  Postoperative pain at 1h, 2 h, 6 h, 24 h, and post-operative days 1 through 5, and at discharge (evaluated with a verbal rating scale (VRS), 0 = no pain, 10 = worst possible pain) until discharge. Pain assessment is performed at rest and during activity (cough).
change in incidence of nausea and vomiting | 1h, 2 h, 24 h post-surgery, and post-operative days 2 through 5, and at discharge from the hospital (approximately 6 days after surgery)
  The incidence of nausea and vomiting at 1h, 2 h, 24 h, and post-operative days 2 through 5, and at discharge from the hospital.

OTHER OUTCOMES:
Time of first bowel movement | After surgery until occurence of first bowel movement during hospital stay (approximately 6 days after surgery)
Time to tolerating liquid intake | After surgery until subject is able to tolerate oral fluids during hospital stay(approximately 6 days after surgery)
Time to tolerating solid intake. | After surgery until subject is able to tolerate solid oral intake during hospital stay (approximately 6 days after surgery)
Postoperative recovery score (QoR-15) | For duration of hospital stay (approximately 6 days after surgery), and 4 weeks after the surgery
  Recovery Scores will be taken at hospital stay (POD 1 to POD 5, Hospital Discharge) and will be repeated at POD 30
6 min Walk Test | For duration of hospital stay (approximately 6 days after surgery), and 4 weeks after the surgery
  If tolerated, individual walks without physical assistance for 6 minutes and the distance is measured. this test will be done at hospital stay (POD 1 to POD 5, Hospital Discharge) and will be repeated at POD 30

CONTACTS AND LOCATIONS:
Overall Officials: Tong J Gan, MD, MHS, Principal Investigator — Duke University; Yang-Sik Shin, MD, Principal Investigator — Shinchon Severance Hospital; Duk-Kyung Kim, MD PhD, Principal Investigator — Samsung Medical Center; Gyu-Jeong Noh, MD PhD, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - Samsung Medical Center, Gangnam-Gu, Seoul
  - Yonsei University College of Medicine, Seodaemun-gu, Seoul
  - Asan Medical Center, Songpa-gu, Seoul